CLINICAL TRIAL: NCT04934085
Title: Impact of Earlier Infection With SARS-COV-2 on Neurological Impairments, Quality of Life, Physical Activity, Social Contacts and Education
Brief Title: COVID-19 Versus Neurological Impairment, Physical Activity, Social Contacts and Education
Status: Completed | Type: Observational
Sponsor: University of Rzeszow (Other)
Responsible Party: Principal Investigator, Agnieszka Guzik, PhD, Principal Investigator, University of Rzeszow
Other Study IDs: COVID-19
Record Dates: First submitted 2021-06-18; First posted 2021-06-22 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Covid19; Neurological Disorder; Balance; Distorted; Gait Disorders, Neurologic; Activity, Motor; Social Isolation; Educational Problems; Quality of Life
MeSH Terms: conditions — COVID-19; Nervous System Diseases; Gait Disorders, Neurologic; Motor Activity; Social Isolation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: subjects who had tested positive and recovered from COVID-19
- Control group: healthy subjects who did not have COVID-19, the controls will be matched to the study group for gender and age

SUMMARY:
The research will make it possible to assess patients who recovered from COVID-19 for the incidence of neurological problems (impaired balance, gait, coordination, concentration and attention), and changes in the quality of life, physical activity, social contacts and education.

DETAILED DESCRIPTION:
The intended size of group - 100 subjects (50 subjects - study group, 50 subjects - control group). The above population was determined based on sample size calculator, with the following parameters: fraction size of 0.9, Confidence Interval of 95%, maximum error of 9%. The proper study will be preceded with a pilot study involving a smaller group of subjects (in order to standardise the surveys, and minimise the relationship between the results of the survey and side-effect factors). After inclusion and exclusion criteria are considered, the subjects will be allocated into two groups:

* study group (subjects who had tested positive and recovered from COVID-19)
* control group (healthy subjects who did not have COVID-19). The controls will be matched to the study group for gender and age.

The examination will be performed once, at the premises of the University of Rzeszów. The participants' condition will be assessed using the following measures:

* static and dynamic balance and risk of falls (force plate and computerised posturography, clinical tests)
* activity in the cerebral cortex of the frontal lobe during focused performance of a task (Hemoencephalography HEG-System)
* concentration and attention, memory and cognitive functions (Bourdon-Wiersma test and Auditory-Verbal Learning Test)
* gait velocity and efficiency (10-meter walk test and 6-minute walk test)
* physical activity (International Physical Activity Questionnaire IPAQ), as well as education, mood, and social contacts (specially designed questionnaire)
* quality of life (SF-36 questionnaire)

ELIGIBILITY:
Inclusion Criteria:

* Informed consent to participate in the study.
* Experienced infection with SARS-COV-2.
* Age 19 - 26 years
* No injuries to lower limbs in the period of 12 months preceding the date of enrolment into the study
* No orthopaedic disorders affecting the lower limbs (including decreased length of the lower limbs)
* No diagnosed neurological diseases or disorders (including labyrinth dysfunction)
* No diagnosed impairment of concentration and attention

Exclusion Criteria:

* Lack of informed consent to participate in the study
* No experience of infection with SARS-COV-2
* Age outside the range of 19 and 27 years
* Confirmed injuries to lower limbs in the period of 12 months preceding the date of enrolment into the study
* Confirmed neurological diseases or disorders, such as impaired balance, concentration and attention.

Ages: 19 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study will be conducted in the population of people living in south-eastern Poland.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Static balance | up to 1 month
  measurements to be performed with a force plate. Centre of Foot Pressure (COP) movements will be assessed in the frontal and sagittal plane (95% confidence ellipse area (COP-area mm2), medium antero-posterior and lateral sway COP (mm), COP average velocity (mm/sec). Stabilographic measurements, each continued for 60 seconds, will be carried out during the following trials: standing on stable ground with eyes open and with eyes closed; standing on unstable ground with eyes open and with eyes closed.
Dynamic balance | up to 1 month
  measurements to be performed using computerised dynamic posturography. The assessment will be performed using Smart EquiTest System from Neurocom. The assessment with take into account delay in response to a destabilising stimulus of mild, moderate and high strength (motor control test - one of the available standard research protocols). The assessment will take into account: Latency - time lapse (in milliseconds) between the onset of support surface translation and the participant's active force response, measured for each limb independently; and Amplitude scaling (or Relative response strength) - strength of the participant's active force response to arrest the angular momentum imparted to the body during the backwards and forwards translations. The response strength will be measured for each leg independently in units of angular momentum (degrees/second) and normalized to body height and weight.
Activity in the cerebral cortex of the frontal lobe | up to 1 month
  measurements to be performed with Hemoencephalography HEG - a system for imaging of cerebral blood oxygenation as well as brain activity. During the examination HEG headset will be placed on the subject's forehead, and any external light stimuli, which could affect the results, will be eliminated. The subject will be required to fully focus on the image displayed on a screen. The examination will comprise a 10-minute session, preceded with one minute test trial during which the indicators will be normalised and the subjects will be prepared for the task. The assessment will take into account HEG ratio mean, max and min. The HEG ratio is: red light (nm) / infrared light (nm)

SECONDARY OUTCOMES:
Concentration and attention | up to 1 month
  measurements to be performed with Bourdon-Wiersma test. During the trial the subject is shown a sheet with a sequence of various letters and digits and he/she is asked to cancel specific letters, e.g., e and r in three minutes. The score reflects the total number of accurately cancelled letters, and a total number of letters omitted or cancelled inaccurately.
Memory and cognitive functions | up to 1 month
  measurements to be performed with Auditory-Verbal Learning Test (AVLT). During the trial the subject is asked to repeat a list of 15 words.
Walking speed | up to 1 month
  measurements to be performed with a 10-meter walk test. During the trials assessing gait velocity (m/s) over a distance of 10 metres, the subjects walk at a self-selected speed.
Walking distance | up to 1 month
  measurements to be performed with a 6-minute walk test. During the trial, the subjects walk at a self-selected speed for 6 minutes.
Self-reliant mobility | up to 1 month
  measurements to be performed with the Timed Up and Go Test. During the trial, the subjects are instructed to get up from a chair with a standard-height backrest and to walk 3 metres, turn round at a specified location, return to the chair and resume the sitting position unassisted
Balance | up to 1 month
  measurements to be performed with Tandem Tests and with a 15-second step test. During Tandem test trials subjects are asked to assume a "tip-top" balance position - the heel of a dominant foot touches the toe of the other with each step. The tasks are used to assess coordination, static and dynamic balance in order to determine the risk of falls. During the 15-second step test, the subject should make as many steps as possible and descend with the entire foot from a 7.5 cm high bench.
Balance and lower limbs muscle strength | up to 1 month
  Measurements to be performed with a sit-to-stand test. During the trial, the subject should perform as many repetitions of standing up and sitting down from a 43.2 cm tall chair in 30 seconds.
Health-related quality of life | up to 1 month
  Measurements to be performed with 20-Item Short Form Survey (SF-20). This questionnaire is a short multi-dimensional instrument that measures six aspects of health status: physical functioning (6 items), role functioning (2 items), social functioning (1 item), mental health (5 items), general health perceptions (5 items), and pain (1 item).
Physical activity level | up to 1 month
  Measurements to be performed with International Physical Activity Questionnaire Short Form (IPAQ-SF). The short form records the "last 7 days recall" activity of four intensity levels: vigorous-intensity activity, moderate-intensity activity, walking, and sitting. Single examination
education, mood, physical activity and social contacts | up to 1 month
  measurements to be performed with a specially designed questionnaire. The self-authored questionnaire consists of questions assessing the impact of Covid-19 pandemic and the related restrictions on the quality of education, knowledge acquisition, frequency and form of physical activity performed, as well as mental state, mood, and changes in social contacts.

CONTACTS AND LOCATIONS:
Overall Officials: Agnieszka Guzik, PhD, Study Chair — University of Rzeszow
Locations (1):
- University of Rzeszów, Rzeszów, Podkarpackie Voivodeship, Poland